CLINICAL TRIAL: NCT04847856
Title: Effectiveness of Diabetic Self-care Education at Primary Health Care Centres in Saudi Arabia: A Pragmatic Randomized Trial in Tabuk
Brief Title: Diabetic Self-care Education at Primary Health Care in Saudi Arabia: A Pragmatic Randomized Trial in Tabuk
Acronym: Diabetescare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tabuk (Other)
Responsible Party: Principal Investigator, Fakhralddin Abbas Mohammed Elfakki, Assistant Professor of Preventive Medicine and Epidemiology, University of Tabuk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-07-TU-077
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Self-care; Preventive Care; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This is a 12 months randomized clustered trial that recruited individuals with type II diabetes mellitus attending primary health care clinics in Tabuk city, Saudi Arabia.
  Health centres will be divided into two groups( intervention& control) using Random Number Generator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- List of health centers that randomly allocated to receive the intervention (Experimental): The intervention was structured Diabetes self-care information, education, and communication (IEC) delivered to the participants at the selected primary health care center level. The Information, education, and communication intervention were delivered by relevant and trained health animators working in chronic care clinics. The intervention was composed of sessions and the participants were planned to attend five structured sessions on diabetes self-care at months: 1, 2, 3,4,5&6. Besides, the participants were provided with a single-page checklist with a to-do list of activities and simple advice that covering the various aspects of diabetes self-care.
  Interventions: Behavioral: Diabetic care Information, education, and communication intervention will be delivered by relevant and trained health animators working in chronic care clinic.
- List of health centers that randomly allocated to receive routine care (No Intervention): The comparators were type II diabetic patients of both genders attending the selected primary health care centres that receiving routinely provided diabetic care including advice from the health care providers. Participants were interviewed at the start of the trial to collect the baseline data about self-care with measurements of blood glucose level, serum cholesterol level, blood pressure, BMI, and waist circumference. At the end of the trial, the sam participants were interviewed to collect end-line data and similar measurements.

INTERVENTIONS:
Behavioral: Diabetic care Information, education, and communication intervention will be delivered by relevant and trained health animators working in chronic care clinic. — The training sessions and the IEC materials were adapted from John Hopkins University studies on self-care for diabetic patients.
  Other Names: Self-care progression card and pictorial IEC messages were prepared and given to the patients or co-family members.
  Arms: List of health centers that randomly allocated to receive the intervention

SUMMARY:
Diabetes Self-care Education (DSCE) is a formal term used to describe the ongoing process of facilitating the knowledge, skills, and ability necessary for diabetes self-care.

Supporting self-care is a crucial aspect of any health service, especially the one that targeting diabetes. It has shown a positive effect on the clinical, psychological, and behavioural aspects of diabetics. However, culturally adapted educational services that recognize the context should be established and used carefully, as most of the social media and YouTube educational products are not relevant most of the time.

Diabetic patients who receive no education about their diabetes, are four times as likely to develop complications as those who do not. Oppositely, those who attending diabetes education programs are less likely to develop long-term complications.

The core question of the trial is to find an answer to the question: how the Diabetes self-care information, education provided by trained health care educator at primary care is effective in controlling patterns of blood glucose, reducing BMI, and enhancing self-care behaviour among diabetic patients attending chronic care clinic compared to the control group receiving routine care for diabetes.

DETAILED DESCRIPTION:
A pragmatic Trial is a modern approach for testing research hypotheses in real life to draw inspiration from the implemented intervention to inform decision making and change in health policy at the level of primary health care and the community.

The trial outcomes could be used in making new policy that directly contributes to the model of care, health economics, and population health management program. It is a 12 months pragmatic randomized trial that will recruit type II diabetic patients attending primary health care centres in Tabuk city.

Conclusion:

Upon successful completion of the trial, the primary and secondary outcomes of the trial like reduction in the blood glucose level, Body Mass Index (BMI), waist circumference, HbA1c, serum cholesterol level, and blood pressure are expected. Besides, the development of new recommendations for diabetes self-care policy, model of care, and on-the-job training at primary health care.

Sample size calculation:

A sample of 250 participants for the two trial arms with an average cluster sample (m) of about 35 participants per cluster is calculated using STATA clustersampsi command. This is by specifying the total number of clusters (k) = 6, the mean for sample1 as (mu1) = 0.6, the mean for sample2 (mu2) = 0.31, the intra-class correlation coefficient (rho) = 0.01, at the power beta (0.8), and significant alpha level of (0.05).

Data analysis:

The collected baseline data and end-line data will be initially analyzed by carrying out both univariate and bivariate analyses. The univariate analysis will summarize data as means, standard deviations while multivariate analysis will yield correlations between the measured variables. Standard statistical tests such as the Student t-test, ANOVA, and F statistic will be used to test for the effects of interventions and to facilitate comparisons between intervention and control groups. Then the data will be further analyzed using multilevel models/hierarchical linear modelling as it allows adjustment of the effect of an intervention for (imbalance on) individual-level and cluster-level baseline predictors of outcomes. The collected data will be analyzed based on the intention to treat evaluate the primary outcomes among both the intervention and control groups i.e. the participants will remain in the group to which they were randomized. Linear regression models will be used for comparing the continuous variables. The BMI as a primary outcome will be analyzed using a linear regression model to find out the effects of the intervention among the intervention groups as well as among the control groups. The secondary outcomes include reduction in blood glucose level, serum cholesterol level, blood pressure, and waist circumference will be analyzed using linear regression models. Statistical significance will be set at 5%.

Missing data will be managed by applying appropriate multiple imputation STAT commands. As the variables are continuous; Markov Chain Monte Carlo (MCMC) method will manage the missing data; it is planned to use SOLA software for managing data (available at http://www.solasmissingdata.com/software.

Generalizability:

This trial is expected to draw some more convenient findings that match the context in Saudi Arabia and other gulf regions. Given the great similarities in sociodemographic, and cultural aspect in addition to the similarities in a health care setting in the whole Kingdom. It is expected that a successful result could fairly be generalized to other health care settings in Saudi Arabia and even to other gulf regions.

Expected limitation:

The quality of data collection is expected to be not to the expected level. This is because the same health provider who will conduct the trial intervention is supposed to carry the data collection task. After all, the physical environment in the health care setting doesn't permit bringing additional staff to complete the task.

Ethical considerations:

Ethical approval will be obtained from the Institutional Review Board in the Faculty of medicine at the University of Tabuk and the Research Ethics Committee at the Ministry of health in Tabuk.

Informed consent: The investigator will make sure that written informed consent is obtained from each participant before randomization and before the participant has undergone any study intervention or data collection procedures. The informed consent will be obtained by the primary health care physician in a special room at the health centre. The primary health care physician will provide the information about the trial and as well ensure that the participant has understood the information. This can be achieved through answering adequately the questions raised by participants; hence, the participants are encouraged to ask questions about the trial and will be given adequate time to decide, voluntarily, either to participate in the trial or not. If a participant needs more to decide, then the primary health care physician should give another appointment for the participants

ELIGIBILITY:
Inclusion Criteria:

* The participants were type II diabetic patients of both genders attending the selected primary health care centers irrespective of their duration of disease and the types of medication currently received. The participants were adults aged 18 years and above.

Exclusion Criteria:

* Children and young adults with juvenile diabetes mellitus were excluded. In addition, severely ill patients, patients with mental disorders were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
To compare the mean differences in the: Blood glucose level, BMI, Waist circumference between intervention and control groups | 12 months
  A reduction in the average blood glucose level, BMI, waist circumference over12 months' duration.

SECONDARY OUTCOMES:
To compare the mean differences in the: HbA1C, Serum cholestrol, and blood pressure between intervention and control groups | 12 months
  A reduction in other biological parameters such as HbA1c, serum cholesterol level, and blood pressure over 12 months' duration.

OTHER OUTCOMES:
To explore the knowlege and skills gained by nurse staff as a result of their participation in the trial intervention. | 12 months
  A qualitative study will be conducted at the end of the project using in-depth interviews with nurse staff who participated in the research to explore the gained knowledge and skills during participation as a secondary outcome, as well.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa K Elnimeiri, MD, Study Chair — Al- Neelain University, Sudan
Locations (1):
- Public Primary Health Care Centers in the Tabuk City, Tabuk, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elfakki FAM, Elnimeiri MK, Assil SM, Frah EA, Abdalla NHI. Effectiveness of diabetes self-care education at primary health care centres in Saudi Arabia: A pragmatic randomized trial in Tabuk. J Family Med Prim Care. 2022 Jan;11(1):144-149. doi: 10.4103/jfmpc.jfmpc_985_21. Epub 2022 Jan 31. PMID 35309655
- See also: Effectiveness of diabetes self-care education at primary health care centres in Saudi Arabia: A pragmatic randomized trial in Tabuk — https://pubmed.ncbi.nlm.nih.gov/35309655/